CLINICAL TRIAL: NCT07323251
Title: Clinical Study on the Effectiveness of Diverse Segments Defocus Optimization in Spectacle Lenses for Slowing Myopia Progression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Mengtian Kang, Principal Investigator, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TREC2024-KY161
Record Dates: First submitted 2025-09-13; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Children With Myopia; Treatment; Multizone Lens Design for Myopic Defocus; Visual Quality; Efficacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Generation of random sequences, determination of random number grouping, and inclusion of subjects by different staff members.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-lens zoning myopia defocus Lens 1 (D.S.D.O) (Experimental)
  Interventions: Device: Diverse Segments Defocus Optimization (D.S.D.O.) spectacle lenses
- Multi-lens zoning myopia defocus Lens 2(D.S.D.O) (Experimental)
  Interventions: Device: Diverse Segments Defocus Optimization (D.S.D.O.) spectacle lenses

INTERVENTIONS:
Device: Diverse Segments Defocus Optimization (D.S.D.O.) spectacle lenses — This clinical trial employs a randomized, parallel-group, superiority design to evaluate two novel optical designs of Diverse Segments Defocus Optimization (D.S.D.O.) myopia management spectacle lenses. A total of 60 myopic Chinese children, aged 6 to 14 years, will be recruited and randomly assigned in a 1:1 ratio to one of two intervention groups. Both groups will receive myopia control spectacles: the Control Group will use D.S.D.O. Lens Design 1, and the Intervention Group will use D.S.D.O. Lens Design 2. Participants are required to wear the assigned spectacles daily for the entire 12-month study duration, except during sleep or other unavoidable circumstances. The spectacles are intended to provide full refractive correction for distance vision while simultaneously incorporating defocus modifications designed to slow myopia progression by manipulating peripheral retinal defocus patterns. The study includes a baseline visit, a dispensing visit, and follow-up assessments at 3, 6, 9

SUMMARY:
Clinical Trial

The goal of this clinical trial is to evaluate the effectiveness of two types of Diverse Segments Defocus Optimization (D.S.D.O.) spectacle lenses in slowing myopia progression in children. It will also assess the safety of these lenses. The main questions it aims to answer are:

Do D.S.D.O. lenses reduce the progression of myopia as measured by changes in cycloplegic refraction and axial length? What adverse events do participants experience when wearing D.S.D.O. lenses? Researchers will compare two optical designs of D.S.D.O. lenses (Intervention Group1: Design 1; Intervention Group2: Design 2) to determine their relative efficacy in controlling myopia progression.

Participants will:

Wear assigned D.S.D.O. lenses daily for 12 months (except during sleep or unavoidable situations).

Attend clinic visits at baseline, 3, 6, 9, and 12 months for comprehensive eye examinations.

Maintain a diary recording daily wear time, visual symptoms, and any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-14 years
* Myopic spherical equivalent refraction between -0.75D and -4.00D (inclusive of -0.75D and -4.00D, based on cycloplegic refraction)
* Astigmatism ≤1.50D
* Anisometropia ≤1.50D
* Best-corrected visual acuity (BCVA) reaching 5.0 (0.00 LogMAR) or better in both eyes; monocular BCVA reaching 5.0 (0.00 LogMAR) or better after wearing myopic defocus spectacles
* Absence of organic ocular diseases
* No history of myopia control treatment within the past three months, including orthokeratology, progressive multifocal lenses, peripheral defocus spectacle lenses, bifocal spectacle lenses, defocus-designed soft hydrophilic contact lenses, other myopia control medications, or light-therapy devices
* Voluntary participation in this clinical study and provision of signed informed consent

Exclusion Criteria:

* History of ocular trauma or surgery
* Systemic diseases affecting visual function
* Inability to cooperate with examinations
* Poor compliance
* Inability to adhere to wearing requirements and follow-up visits during the trial period

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Spherical Equivalent Refraction (SER) | From enrollment to the end of treatment at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China